CLINICAL TRIAL: NCT05422027
Title: Selinexor(ATG-010) Plus Bortezomib, Lenalidomide and Dexamethasone (XVRd) in High Risk Newly Diagnosed Multiple Myeloma
Brief Title: Selinexor Plus VRd in High Risk Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xia Zhongjun (Other)
Collaborators: Antengene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Xia Zhongjun, Chief physician, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-010-IIT-MM-005
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
Keywords: Selinexor; ATG-010; Newly Diagnosed; High Risk
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; Bortezomib; Lenalidomide; Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Selinexor-VRd（XVRd） (Experimental): bortezomib SC 1.3mg/sqm on day 1,4,8,11, lenalidomide oral 25 mg on day 1-14, and dexamethasone 40mg on day 1,8,15 in a 21-day cycle; Selinexor dose escalation: 40，60mg respectively on day 1,8,15 for 21-days cycles. Then Selinexor will be given at the recommended dose level on phase II.
  Interventions: Drug: Selinexor; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Selinexor (ATG-010# is a first-in-class, oral selective exportin 1 (XPO1) inhibitor (1,2). Selinexor functions by binding with and inhibiting the nuclear export protein XPO1 (also called CRM1), leading to the accumulation of tumor suppressor proteins in the cell nucleus along with inhibition of translation of oncoprotein mRNAs.
  Selinexor dose escalation: 40, 60mg respectively on day 1,8,15 for 21 days cycles
  Other Names: ATG-010; Xpovio
Drug: Bortezomib — The investigators gave patients subcutaneous bortezomib 1.3mg/sqm on days 1, 8,15 of a 21- day cycle.
  standard bortezomib-lenalidomide-dexamethasone
  Other Names: Velcade
Drug: Lenalidomide — The investigators gave patients oral lenalidomide 25mg on days 1 to 14 of a 21-day cycle.
  standard bortezomib-lenalidomide-dexamethasone
  Other Names: Revlimid
Drug: Dexamethasone — The investigators gave patients oral dexamethasone 40mg on days 1, 8, 15 of a 21-day cycle.
  standard bortezomib-lenalidomide-dexamethasone
  Other Names: Dexamethasone Acetate

SUMMARY:
This is a single-arm and open-label study to explore XVRd (ATG-010, Bortezomib, Lenalidomide and Dexamethasone) regimen in high-risk newly diagnosed multiple myeloma.The primary objective of the dose escalation study is to determine the safety, tolerability, and recommended phase II dose (RP2D) of selinexor; Then dose expansion at the RP2D level based on dose escalation phase will be conducted to evaluate the efficacy, safety and tolerability.The enrollment period for this study is expected to be approximately 12 months.

The study will end when all patients have completed 12 cycles treatment/follow-up since the initiation of the study drug, or the last patient has expired, has been lost to follow-up, or has withdrawn consent, whichever occurs first.

DETAILED DESCRIPTION:
This is a single-arm and open-label study to explore XVRd (ATG-010, Bortezomib, Lenalidomide and Dexamethasone) regimen in high-risk newly diagnosed multiple myeloma. Approximately 3-42 patients will be enrolled in the study. In dose escalation phase, patients with high-risk NDMM will be treated with VRd standard regimen (bortezomib 1.3mg/m2 SC on day1,4,8,11, lenalidomide 25 mg on day 1-14 and dexamethasone 40mg on day 1,8,15 in a 21-day cycle) plus escalating doses of selinexor 40 mg or 60 mg on days 1, 8, and 15 of each cycle in a 3+3 design. The primary objective of the dose escalation study is to determine the safety, tolerability,and recommended phase II dose (RP2D) of selinexor; Then dose expansion at the RP2D level based on dose escalation phase will be conducted to evaluate the efficacy, safety and tolerability. All of the patients will receive 12 cycles of XVRd , and subjects can choose maintenance treatment with XR after 12 cycles of XVRd.The primary objective of the dose escalation study is to determine the safety, tolerability, and recommended phase II dose (RP2D) of selinexor; Then dose expansion at the RP2D level based on dose escalation phase will be conducted to evaluate the efficacy, safety and tolerability.

The enrollment period for this study is expected to be approximately 12 months. The study will end when all patients have completed 12 cycles treatment/follow-up since the initiation of the study drug, or the last patient has expired, has been lost to follow-up, or has withdrawn consent, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible to enroll in this study:

  1. Willing and able to written informed consent (ICF) .
  2. Age ≥ 18 years.
  3. Newly diagnosed multiple myeloma as defined by IMWG(Rajkumar, Dimopoulos et al. 2014) , measurable disease as defined IMWG 2016 criteria(Table 5) (Kumar, Paiva et al.2016), and meet at least one of the following criteria:

     1. Serum M-protein (SPEP) ≥ 5 g/L, If the MM type is IgA/IgD, that can be substituted by IgA/IgD quantitative level.
     2. 24 hours-Urinary M-protein excretion ≥ 0.2 g (200 mg)
     3. Serum FLC ≥ 100 mg/L with abnormal FLC ratio ( FLC Normal ratio:0.26 to 1.65)
  4. According to mSMART 3.0 definition for high risk multiple myeloma:

     1. High Risk genetic Abnormalities t(4;14) , t(14;16) , t(14;20) , Del 17p, p53 mutation, Gain 1q
     2. R-ISS Stage 3
     3. High Plasma Cell S-phase
     4. GEP: High risk signature
  5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2. ECOG PS 3 allowed, if caused by myeloma.
  6. Patients must have received no prior chemotherapy for multiple myeloma. Patients must have received no prior radiotherapy to a large area of the pelvis (more than half of the pelvis). Patients must have received no prior steroid treatment for myeloma with the exception of a maximum of 14 days of treatment for symptom control.
  7. Adequate hepatic function: total bilirubin < 1.5× upper limit of normal (ULN) (for patients with Gilbert's syndrome, a total bilirubin of < 3× ULN is required), AST < 2× ULN, and ALT < 2× ULN.
  8. Adequate renal function: estimated creatinine clearance ≥ 30 mL/min (calculated using the formula of Cockroft-Gault).
  9. Adequate hematopoietic function within 7 days prior to C1D1 and met the following criteria: White blood cell (WBC) count ≥1.5×109/L, Absolute neutrophil count (ANC)≥1.0×109/L, Hemoglobin (HB) ≥85g/L and Platelet count (PLT) ≥75×109/L (patients whom <50% of bone marrow nucleated cells are plasma cells) or PLT ≥ 50×109/L (patients whom ≥ 50% of bone marrow nucleated cells are plasma cells).
  10. Patients could not receive hematopoietic growth factor treatment within 2 weeks prior to screening, These growth factors include Erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), Granulocyte macrophages-colony stimulating factor (GM-CSF), Platelet agonist, etc (Eltrombopag, Thrombopoietin (TPO), Interleukin-11).
  11. Patients receive transfusions of blood products:

      1. At least 2 weeks elapsed between the screening hemoglobin assessment and the last red blood cell infusion,
      2. And at least 1 week elapsed between the screening platelet assessment and the last platelet infusion.
  12. Patients must be able to take prophylactic anticoagulant therapy as recommended by the study.
  13. Female patients of childbearing potential must meet below two criteria:

      1. must agree to use effective contraception methods since signature in ICF, throughout the study and for 3 months following the last dose of study treatment.
      2. must have a negative serum pregnancy test at screening. Note: A woman is considered of childbearing potential following menarche and until becoming postmenopausal (defined as no menstrual period for a minimum of 12 months) or permanently sterile (having undergone a hysterectomy, bilateral salpingectomy or bilateral oophorectomy). A woman who is taking oral contraceptive or using intrauterine device is considered of childbearing potential.

Male patients (including those who have received vasectomy) must use a condom if sexually active with a female of child-bearing potential throughout the study and for 3 months following the last dose of study treatment.

Exclusion Criteria:

* Patients who meet any of the following criteria will not be enrolled:

  1. Plasma cell leukemia.
  2. Documented active amyloidosis.
  3. Involvement of the central nervous system(CNS) by Multiple myeloma.
  4. Prior exposure to a SINE compound, including ATG-010.
  5. Currently, whether or not the patient is on medication, > Grade 2 peripheral neuropathy or ≥ Grade ≥ 2 painful neuropathy at baseline.
  6. Known intolerance, hypersensitivity, or contraindication to glucocorticoids, bortezomib, lenalidomide, and Selinexor (ATG-010) .
  7. Active, unstable cardiovascular function, as indicated by the presence of:

     1. Symptomatic ischemia, or
     2. Uncontrolled clinically significant conduction abnormalities (eg, patients with ventricular tachycardia on anti-arrhythmics are excluded; patients with first degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), or
     3. Congestive heart failure of New York Heart Association Class ≥3 or known left ventricular ejection fraction <40%, or
     4. Myocardial infarction within 6 months prior to C1D1.
  8. Known positive serology for HIV or HIV seropositivity.
  9. Known active hepatitis A, B, or C infection; eg. positive for HCV RNA or HBV-DNA.
  10. Women who are pregnant or nursing.
  11. Life expectancy of less than 6 months.
  12. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
  13. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
  14. Contraindication to any of the required concomitant drugs or supportive treatments.
  15. Has any concurrent diseases or complications that is likely to interfere with the study procedures.
  16. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Maximum Tolerated Dose (MTD) | Assessed from the date of first dose of study treatment to the first cycle ends (maximum 21days) ;
  The MTD will be determined by study definition as the highest dose level without significant safety and tolerability concern.
Dose Escalation: Recommended Phase 2 Does (RP2D) | Assessed from the date of first dose of study treatment to the first cycle ends (maximum 21days) ;
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for the dose expansion arms, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation portion of the study.
Dose Expansion: MRD negative remission | At any time up to 12 months after XVRD treatment
  MRD negative remission (<10-5) as defined by IMWG consensus

SECONDARY OUTCOMES:
complete response (CR) | Cycle 1 Day 1 (each cycle consists of maximum 21 days) until a VGPR, CR or PR (up to 12 cycles)
  complete response (CR) and stringent complete response (sCR)
Overall Survival (OS) | 12 months
  Occurrence of death regardless of cause
Progression-Free Survival (PFS) | 12 months
  Duration from start of study treatment to PD or death (regardless of cause), whichever comes first
Duration of Response (DOR) | 12 months
  Duration from the first observation of at least PR to time of disease progression, or deaths due to disease progression, whichever occurs first
Clinical Benefit Rate (CBR) | 12 months
  Clinical Benefit Rate (CBR=ORR+Minor Response [MR])
Disease Control Rate (DCR) | 12 months
  Disease Control Rate (DCR=CBR+Stable Disease[SD; for a minimum of 12 weeks])
Number of Participants with Adverse Events | From first dose of study drug administration to end of treatment (up to 12 months)
  Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongjun Xia, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (4):
- China (4):
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center; State Key Laboratory of Oncology in South China,, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
All IPD results are used for publication,and can be shared with other investigators and sponsors
Supporting Information: Study Protocol
Time Frame: Study Protocol can be shared Starting 12 months after publication
Access Criteria: Study Protocol must not be shared with non-participants until after publication and must be authorized by the principal investigator and sponsors